CLINICAL TRIAL: NCT04028297
Title: Focus Cardiac Ultrasound in Patients With Undifferentiated Shock: Prospective Observational Study
Brief Title: Focus Cardiac Ultrasound in Patients With Shock
Acronym: echoshock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-035
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Shock
Keywords: Shock; emergency; undifferentiated; ultrasound
MeSH Terms: conditions — Shock; Emergencies; Disorders of Sex Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Focus cardiac ultrasound (FoCUS)

SUMMARY:
The aim of this study is to analyze in patients with undifferentiated shock, the concordance of initial treatment before and after Focus cardiac ultrasound (FoCUS) in comparison with the reference one established by an adjudication committee

DETAILED DESCRIPTION:
Focus cardiac ultrasound (FoCUS) has already demonstrated its ability to reduce diagnosis uncertainty in patients with undifferentiated shock. However, adequacy of initial treatment has not been investigated.

In patients with undifferentiated shock, after clinical evaluation, the physician states its hypothesis and initial treatment intention in closed list. He realizes a FoCUS, states another time the hypothesis and begins treatment according to FoCUS results. An adjudication committee with all the patient's file will state the reference hypothesis and treatment

ELIGIBILITY:
Inclusion Criteria:

* Undifferentiated shock defined by systolic arterial pressure < 90 mm Hg

Exclusion Criteria:

* hemorrhagic shock
* cardiac arrest
* anaphylactic shock
* documented end-of-life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with undifferentiated shock in the Emergency Department
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
concordance of initial treatment after FoCUS with Kappa coefficient | Hospitalization duration, up to one month
  concordance between initial treatment after clinical procedure, after FoCUS in comparison with the reference stated by the adjudication committee with Kappa coefficient

SECONDARY OUTCOMES:
duration of FoCUS | Hospitalization duration, up to one month
  concordance between initial diagnosis after clinical procedure, after FoCUS in comparison with the reference stated by the adjudication committee
difficulty of FoCUS | Hospitalization duration, up to one month
  concordance between initial diagnosis after clinical procedure, after FoCUS in comparison with the reference stated by the adjudication committee

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No